CLINICAL TRIAL: NCT06716307
Title: Comparing the Pharmacokinetics of Cagrilintide and Semaglutide Following Single Subcutaneous Doses of Different CagriSema Presentations, in a Crossover Manner in Adult Participants With Overweight or Obesity
Brief Title: A Research Study to Compare Blood Levels of Cagrilintide and Semaglutide After Single Doses of Different Versions of Injectable CagriSema in Adults With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-8259; U1111-1309-7476 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence 1 (Experimental): Participants will receive a single subcutaneous (s.c.) dose of CagriSema (cagrilintide B and semaglutide I) in DV3384 pen-injector in period 1 followed by a single s.c. dose of CagriSema A in PDS290 pen-injector in period 2 separated by a wash out period of minimum 7 weeks.
  Interventions: Drug: CagriSema (cagrilintide B and semaglutide I); Drug: CagriSema A
- Treatment sequence 2 (Experimental): Participants will receive a single s.c. dose of CagriSema A in PDS290 pen-injector in period 1 followed by a single s.c. dose of CagriSema (cagrilintide B and semaglutide I) in DV3384 pen-injector in period 2 separated by a wash out period of minimum 7 weeks.
  Interventions: Drug: CagriSema (cagrilintide B and semaglutide I); Drug: CagriSema A

INTERVENTIONS:
Drug: CagriSema (cagrilintide B and semaglutide I) — Cagrilintide and semaglutide will be administered subcutaneously using DV3384 pen-injector.
Drug: CagriSema A — Cagrilintide and semaglutide will be administered subcutaneously using PDS290 pen-injector.

SUMMARY:
This study will compare the blood levels of cagrilintide and semaglutide when the same dose is given in two different versions of CagriSema. CagriSema is a medicine that combines two medicines called cagrilintide and semaglutide. It is still being tested in studies and is not yet available for doctors to prescribe. Participants will get an injection with each of the two versions of CagriSema at two different times at the clinic. Like all medicines, the study medicine may have side effects. The study will last for about 18 weeks.

ELIGIBILITY:
Inclusion criteria:

* Male or female.
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) between 27.0 and 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.

Overweight should be due to excess adipose tissue, as judged by the investigator.

- Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Previous dosing with an amylin analogue.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* Glycosylated haemoglobin (HbA1c) greater than or equal to (>=) 6.5 percent (48 millimoles per mole [mmol/mol]) at screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,cagri,0.25 milligram (mg)/0.25mg,SD: Area under the cagrilintide concentration-time curve after a single dose 0.25 mg/0.25 mg CagriSema A in PDS290 pen-injector or CagriSema in DV3384 pen-injector | From 0 hours (pre-dose) to 1176 hours (post-dose)
  Measured in hours*nanomoles per liter (h*nmol/L).
Cmax,cagri,0.25mg/0.25mg,SD: Maximum concentration of cagrilintide after a single dose 0.25 mg/0.25 mg CagriSema A in PDS290 pen-injector or CagriSema in DV3384 pen-injector | From 0 hours (pre-dose) to 1176 hours (post-dose)
  Measured in nanomoles per liter (nmol/L).
AUC0-∞,sema,0.25mg/0.25mg,SD: Area under the semaglutide concentration-time curve after a single dose 0.25 mg/0.25 mg CagriSema A in PDS290 pen-injector or CagriSema in DV3384 pen-injector | From 0 hours (pre-dose) to 1176 hours (post-dose)
  Measured in h*nmol/L.
Cmax,sema,0.25mg/0.25mg,SD: Maximum concentration of semaglutide after a single dose 0.25 mg/0.25 mg CagriSema A in PDS290 pen-injector or CagriSema in DV3384 pen-injector | From 0 hours (pre-dose) to 1176 hours (post-dose)
  Measured in nmol/L.

SECONDARY OUTCOMES:
Number of adverse events | From first investigational medicinal product (IMP) administration (Day 1) to the end of study visit (Day 99)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Celerion, Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com